CLINICAL TRIAL: NCT03103854
Title: The Impact of Novel Strategies to Improve Cardiometabolic Status and Adherence to Exercise Regimens in Patients at High Risk for Cardiovascular Disease
Brief Title: Novel Strategies to Improve Cardiometabolic Status and Adherence to Exercise Regimens in Patients at High Risk for Cardiovascular Disease
Acronym: BURST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge Cardiac Care Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CCCBE1418
Record Dates: First submitted 2017-03-28; First posted 2017-04-06 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 2; Myocardial Infarction; Coronary Artery Disease; Atrial Fibrillation; Congestive Heart Failure
Keywords: Exercise; Secondary Prevention; Diabetes; Rehabilitation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocardial Infarction; Coronary Artery Disease; Atrial Fibrillation; Heart Failure; Motor Activity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is a 2x2 of burst physical activity (BURST) vs moderate intensity continuous training (MICT) and text message reminders vs no text message reminders. Patients will be randomized to either BURST or MICT and then further randomized to either receive text message reminders or not receive text message reminders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): Patients in the "Control" arm of the study performed Moderate Intensity Continuous Training (MICT) and did not receive text message reminders.
  Interventions: Behavioral: Moderate Intensity Continuous Training
- BURST (Experimental): Patients in the "BURST" arm of the study performed BURST physical activity and did not receive text message reminders
  Interventions: Behavioral: BURST physical activity
- Text Message Reminders (Experimental): Patients in the "Text Message Reminders" arm of the study performed Moderate Intensity Continuous Training and received text message reminders.
  Interventions: Behavioral: Text Message Reminders; Behavioral: Moderate Intensity Continuous Training
- BURST and Text Message Reminders (Experimental): Patients in the "BURST and Text Message Reminders" arm of the study performed Burst physical activity and received text message reminders
  Interventions: Behavioral: BURST physical activity; Behavioral: Text Message Reminders

INTERVENTIONS:
Behavioral: BURST physical activity — BURST is a novel exercise regimen consisting of three daily periods of 10 minutes of high intensity physical activity spread throughout the day.
  Other Names: Exercise Snacks
  Arms: BURST; BURST and Text Message Reminders
Behavioral: Text Message Reminders — Patients were sent daily text message reminders to remind them to exercise.
  Arms: BURST and Text Message Reminders; Text Message Reminders
Behavioral: Moderate Intensity Continuous Training — This is the current standard of care for cardiac rehabilitation patients. It consists of 1 daily period of 30 minutes of moderate intensity physical activity.
  Other Names: MICT
  Arms: Control; Text Message Reminders

SUMMARY:
This is a 2x2 study examining the impacts of a novel exercise regimen and daily text message reminders in patients at high risk for cardiovascular disease. Patients participating in cardiac rehabilitation will be randomized to either moderate intensity continuous training (MICT) or a novel exercise regimen consisting of three periods of high intensity exercise, called BURST exercise. Additionally, half of the patients in each exercise group will be randomized to receive daily text message reminders to improve adherence to the prescribed exercise regimen.

DETAILED DESCRIPTION:
Numerous studies have demonstrated the important cardiometabolic impacts of high intensity exercise in patients at high risk for cardiovascular disease. It is also known that adherence to exercise regimens is poor within these populations. This study compares the impacts of the current standard of care, moderate intensity continuous training (MICT) to a novel exercise regimen called BURST exercise within a population of patients at high risk for cardiovascular disease. BURST exercise consists of three periods of high intensity physical activity spread throughout the day. Additionally, as mobile technologies continue to be used more to improve adherence to exercise regimens, this study also seeks to compare the impacts of text message reminders in patients prescribed each of the exercise regimens examined in this study. Thus, patients were also randomized to either receive daily text message reminders, or to receive no text message reminders.

Recruitment will be conducted at Cambridge Cardiac Rehab in Ontario, Canada. Potential study subjects are evaluated for inclusion and exclusion criteria, give written informed consent, and are randomized, in a 1:1 ratio, to either MICT or BURST exercise. Additionally, patients are then randomized in a 1:1 ratio to either receive text message reminders or not receive text message reminders.

Patients prescribed the MICT regimen will be asked to exercise for 30 minutes per day at moderate intensity, at least five days per week. Patients prescribed the BURST exercise regimen will be asked to exercise for 10 minutes per session, three times a day at high intensity, at least five days per week. Patients randomized to receive text message reminders will be sent four daily text message reminders reading: "Please remember to exercise for 30 minutes today."

Adherence to exercise regimens will be measured by daily logbooks. Patients are asked to log the times they exercised and for what duration. BRUCE protocol stress tests will be conducted for all patients at baseline (before beginning the study), after three months and after one year. Hemoglobin A1C blood tests, height and weight measurements and lipid profile blood tests will also be conducted at baseline (before the beginning of the study), after three months and after one year.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetic patients (within the last 3 months)
* Participating in on-site the diabetes rehabilitation program at Cambridge Cardiac Rehab
* Deemed capable of high-intensity exercise

Exclusion Criteria:

* Known or suspected cardiovascular disease
* Diabetic end-organ damage
* Cerebrovascular disease
* Peripheral vascular disease
* Arthritis
* Joint disease
* Taking anti-glycemic medications
* Taking lipid lowering medications
* Ischemia, hypoxia, arrhythmia or hemodynamic instability during a stress test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1C at 12 months | 12 months
  Hemoglobin A1C blood test

SECONDARY OUTCOMES:
LDL at 3 months | 3 months
  Calculated Low Density Lipoprotein from blood tests
LDL at 12 months | 12 months
  Calculated Low Density Lipoprotein from blood tests
HDL at 3 months | 3 months
  Measured High Density Lipoprotein from blood tests
HDL at 12 months | 12 months
  Measured High Density Lipoprotein from blood tests
Triglycerides at 3 months | 3 months
  Measured Triglycerides from blood tests
Triglycerides at 12 months | 12 months
  Measured Triglycerides from blood tests
BMI at 3 months | 3 months
  Calculated Body Mass Index based on height and weight measurements
BMI at 12 months | 12 months
  Calculated Body Mass Index based on height and weight measurements
Exercise Capacity at 3 months | 3 months
  Timed number of minutes achieved on a Bruce Protocol treadmill stress test
Exercise Capacity at 12 months | 12 months
  Timed number of minutes achieved on a Bruce Protocol treadmill stress test
Monthly Duration of Exercise | Months 1-12
  Average number of minutes of exercise logged by patients in daily logbooks
HbA1C at 3 months | 3 months
  Hemoglobin A1C blood test

CONTACTS AND LOCATIONS:
Overall Officials: Avinash Pandey, Principal Investigator — Western University, Canada
Locations (1):
- Cambridge Cardiac Rehab, Cambridge, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaede P, Lund-Andersen H, Parving HH, Pedersen O. Effect of a multifactorial intervention on mortality in type 2 diabetes. N Engl J Med. 2008 Feb 7;358(6):580-91. doi: 10.1056/NEJMoa0706245. PMID 18256393
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Armstrong MJ, Sigal RJ, Arena R, Hauer TL, Austford LD, Aggarwal S, Stone JA, Martin BJ. Cardiac rehabilitation completion is associated with reduced mortality in patients with diabetes and coronary artery disease. Diabetologia. 2015 Apr;58(4):691-8. doi: 10.1007/s00125-015-3491-1. Epub 2015 Jan 26. PMID 25742772
- [Background] Francois ME, Little JP. Effectiveness and safety of high-intensity interval training in patients with type 2 diabetes. Diabetes Spectr. 2015 Jan;28(1):39-44. doi: 10.2337/diaspect.28.1.39. PMID 25717277
- [Background] Thakkar J, Kurup R, Laba TL, Santo K, Thiagalingam A, Rodgers A, Woodward M, Redfern J, Chow CK. Mobile Telephone Text Messaging for Medication Adherence in Chronic Disease: A Meta-analysis. JAMA Intern Med. 2016 Mar;176(3):340-9. doi: 10.1001/jamainternmed.2015.7667. PMID 26831740